CLINICAL TRIAL: NCT02519738
Title: Granulation Tissue at G Tube Site: Treatment With Kenalog vs Chemical Cauterization With Silver Nitrate vs Soap Washcloth Abrasion
Brief Title: Granulation Tissue Treatment: Silver Nitrate vs Kenalog vs Washcloth Abrasion
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: enrollment difficulties
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ronald Bruce Hirschl, MD, Professor of Pediatric Surgery & Head, Department of Pediatric Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00077762
Record Dates: First submitted 2015-07-22; First posted 2015-08-11 (Estimated); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Other Abnormal Granulation Tissue Nos
MeSH Terms: interventions — Silver Nitrate; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Silver Nitrate (Active Comparator): Silver Nitrate is supplied in the form of pre-packaged applicator sticks to parents and patients. The concentration is 75% Silver Nitrate and 25% Potassium Nitrate. Application will be done 3 times a week for a period of 3 weeks.
  Interventions: Drug: Silver Nitrate
- Kenalog (Triamcinolone) (Active Comparator): Kenalog is a topical corticosteroid that shares anti-inflammatory, anti-pruritic, and vasoconstrictive actions.The dosage of Kenalog used in the study is 0.5%. Application is topical, and the frequency is 3 times a day for the 3 week trial period. FDA approved use of Kenalog in the treatment of inflammatory and pruritic manifestations of corticosteroid-responsive dermatoses. It has not been studied whether Kenalog has any proven advantage over Silver nitrate in the treatment of granulation tissue, but it has been used for the treatment of granulation tissue at the gastrostomy site with good effect.
  Interventions: Drug: Kenalog (Triamcinolone)
- Washcloth Abrasion (Active Comparator): Washcloth abrasion will be done with regular soap and water applied to a washcloth. The granulation tissue will be gently washed and abraded once daily for three weeks.
  Interventions: Other: Washcloth Abrasion

INTERVENTIONS:
Drug: Silver Nitrate — Silver nitrate to be applied 3 times weekly for a period of 3 weeks.
  Arms: Silver Nitrate
Drug: Kenalog (Triamcinolone) — Triamcinolone will be applied as an ointment to the granulation tissue site three times daily for a total of three weeks.
  Arms: Kenalog (Triamcinolone)
Other: Washcloth Abrasion — Gentle wash and abrasion with washcloth done once daily for a total of 3 weeks.
  Arms: Washcloth Abrasion

SUMMARY:
Granulation tissue, or excess tissue, forms around gastrostomy tube sites and is a common problem seen in the pediatric surgery population. There is no standard treatment that has been identified in clinical practice to treat granulation tissue effectively. Clinicians prescribe treatments of varying nature to help treat this condition. By conducting this study, the investigators hope to identify if there is any difference in the treatment groups and if there is any superiority for one treatment over the other. The three arms in the study are Silver Nitrate treatment, treatment with Kenalog, and Washcloth abrasion. Treatments will continue over a period of three weeks, and the progress will be followed using surveys and photographs.

DETAILED DESCRIPTION:
Hypergranulation tissue surrounding gastrostomy tube sites in pediatric patients is a significant problem. This tissue may cause drainage or bleeding that bothers patients and parents. Numerous methods of treatment are used for treatment of hypergranulation tissue, but no data exists to support one method of treatment over another. The investigators plan to perform a prospective randomized trial of three different therapies (silver nitrate cauterization, topical kenalog, and soap cloth abrasion) to identify the best treatment modality. Participants will be followed via office visit at four and eight weeks after initiation of therapy. Measurements of the granulation tissue and photographs will be obtained pre treatment and at each post treatment visit. In addition parents will be asked to fill out a pre and post treatment survey regarding improvement in symptoms. Investigators plan to enroll 120 patients total with the intention of having 40 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* Any patient falling within age group with granulation tissue around G tube site

Exclusion Criteria:

* Patients falling outside of age group range

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B Hirschl, MD, Principal Investigator — Univeristy of Michigan
Locations (1):
- C.S. Mott Children's Hospital, University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Silver Nitrate | Kenalog (Triamcinolone) | Washcloth Abrasion
Started | 20 | 17 | 15
Completed | 6 | 4 | 3
Not Completed | 14 | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silver Nitrate | Kenalog (Triamcinolone) | Washcloth Abrasion | Total
Number analyzed (Participants) | 20 | 17 | 15 | 52
Age, Customized [Mean (Full Range); unit: years]
  Age in years | 5.38 [.25 to 16] | 3.39 [.42 to 8] | 6.47 [.58 to 17] | 5.04 [.25 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 8 | 20
  Male | 14 | 11 | 7 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 0 | 6
  White | 12 | 11 | 13 | 36
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 15 | 52

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Size (mm) of Granulation Tissue
Description: Measurements are calculated from photographs taken with a millimeter ruler next to granulation tissue on a horizontal plane and a vertical plane. The horizontal and vertical diameters are averaged and then halved, to give a radius which is squared and multiplied by Pi for an approximate area. The area at 8 weeks is subtracted from the area at baseline, to calculate the change and then they are averaged across the individuals with pre and post data for the arm. This approximation is limited by the fact that the shape and all the dimensions of the granulation tissue are highly variable. In order to measure the change the horizontal and vertical diameters were averaged as if they were a circle. This is a limitation of the analysis.
Time Frame: 8 weeks
Population: Population consists of those participants for whom pre and 8 week data is available.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Silver Nitrate | Kenalog (Triamcinolone) | Washcloth Abrasion
Number analyzed (Participants) | 7 | 4 | 4
mm^2
  Pre-Treatment | 101.12 (138.60) | 83.14 (13.08) | 121.72 (71.26)
  Post-Treatment | 22.36 (52.94) | 45.06 (21) | 140.54 (96.51)
  Change from pre-post | 78.77 (149.10) | 37.95 (31.62) | -18.81 (106.58)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Silver Nitrate | Kenalog (Triamcinolone) | Washcloth Abrasion
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/17 | 1/15
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 1/15
Other Adverse Events (participants affected / at risk) | 6/20 | 4/17 | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Silver Nitrate (N=20) | Kenalog (Triamcinolone) (N=17) | Washcloth Abrasion (N=15)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 — Inflammation and drainage around g-tube site; hospitalized for neutropenia/fever and cellulitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Silver Nitrate (N=20) | Kenalog (Triamcinolone) (N=17) | Washcloth Abrasion (N=15)
Pain with Rx/burning (Skin and subcutaneous tissue disorders) | 4 | 1 | 1
bleeding at site (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
abscess at site (Infections and infestations) | 0 | 0 | 1
worsening granulation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
infection at G tube site (Infections and infestations) | 0 | 1 | 0
irritation/inflammation at G tube site (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
dislodged G tube (Injury, poisoning and procedural complications) | 1 | 0 | 0 — and esophageal biopsy

LIMITATIONS AND CAVEATS:
Because evaluable data was less than 1/4 of what was sought, no statistical power was achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT02519738/Prot_SAP_000.pdf